CLINICAL TRIAL: NCT04324905
Title: A Randomized, Open-label, Multiple Dose, Crossover Study to Compare the Safety, Pharmacokinetics and Pharmacodynamics of HIP1802 to HGP1705 in Healthy Volunteers
Brief Title: Study to Compare the Safety, Pharmacokinetics and Pharmacodynamics of HIP1802 to HGP1705 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-ESOB-101
Record Dates: First submitted 2020-02-28; First posted 2020-03-27 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental)
  Interventions: Drug: HIP1802; Drug: HGP1705
- Sequence 2 (Experimental)
  Interventions: Drug: HIP1802; Drug: HGP1705

INTERVENTIONS:
Drug: HIP1802 — Test drug
Drug: HGP1705 — Reference drug

SUMMARY:
A Phase 1 Study to Compare the Safety, Pharmacokinetics and Pharmacodynamics of HIP1802 to HGP1705 in Healthy Volunteers

DETAILED DESCRIPTION:
A Randomized, Open-label, Multiple dose, Crossover Study to Compare the Safety, Pharmacokinetics and Pharmacodynamics of HIP1802 to HGP1705 in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers in the age between 19 and 50 years old.
* Body mass index (BMI) in the range of 19 to 28 kg/m2 and weight 55.0kg to 90.0kg.
* After fully hearing and understanding the details of this clinical trial, Subjects who have willingness to sign of informed consent before the screening.
* Subject who are eligible from physical examination, clinical laboratory test by investigators judgment.

Exclusion Criteria:

* Gastrointestinal disorders (gastrointestinal ulcers, gastritis, stomach cramps, gastro-esophageal reflux disease, Crohn's disease or chronic pancreatitis) or gastrointestinal surgery (except for simple cecal or hernia surgery) which may affect the safety and pharmacokinetic evaluation of test drug.
* Subjects who have a history of hypersensitivity or clinically significant hypersensitivity to investigational product or the same component or other drugs (aspirin, antibiotics, etc.).
* Aspartate aminotransferase and alanine aminotransferase exceed 1.5 times the upper limit of normal range from screening laboratory results before randomization.
* Subject who continues to drink (21 units / week, 1 unit = 10 g of pure alcohol) within a month before the screening visit or who cannot abstain during the hospital stay.
* Heavy smoker (>10 cigarettes/day).

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
AUClast | 0-24hours
Reduced rate from baseline in 24h integrated gastric pH | 0-24hours

SECONDARY OUTCOMES:
Cmax | 0-24hours
Tmax | 0-24hours
t1/2 | 0-24hours
CL/F | 0-24hours
Vd/F | 0-24hours
AUCtau | 0-24hours
Cmin,ss | 0-24hours
Cmax,ss | 0-24hours
t1/2,ss | 0-24hours
CLss/F | 0-24hours
Vd,ss/F | 0-24hours
Reduced rate from baseline in 24h integrated gastric pH | 0-24hours
Duration time with integrated gastric pH>4 / 24hr | 0-24hours
Median 24 hr gastric pH | 0-24hours

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim Y, Bae S, Jeon I, Kwon J, Hong SH, Kim NY, Yu KS, Jang IJ, Lee S. Pharmacokinetics and Pharmacodynamics of a Fixed-Dose Combination of Esomeprazole and Magnesium Hydroxide Compared to the Enteric-Coated Esomeprazole. Clin Ther. 2024 Nov;46(11):870-876. doi: 10.1016/j.clinthera.2024.08.006. Epub 2024 Sep 16. PMID 39289057